CLINICAL TRIAL: NCT01034982
Title: A Phase I Open-label, Single-centre, Two Cohort Crossover Study to Assess the Relative Bioavailability After Oral Administration of AZD9668 Free Base Dosed as a Suspension Compared to AZD9669 Tosylate Salt Dosed as a Tablet
Brief Title: AZD9668 Relative Bioavailability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: D0520C00017
Record Dates: First submitted 2009-12-14; First posted 2009-12-18 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — N-((5-(methanesulfonyl)pyridin-2-yl)methyl)-6-methyl-5-(1-methyl-1H-pyrazol-5-yl)-2-oxo-1-(3-(trifluoromethyl)phenyl)-1,2-dihydropyridine-3-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): tosylate salt tablet
  Interventions: Drug: AZD9668
- 2 (Experimental): free suspension
  Interventions: Drug: AZD9668
- 3 (Experimental): tosylate salt tablet
  Interventions: Drug: AZD9668
- 4 (Experimental): free suspension
  Interventions: Drug: AZD9668

INTERVENTIONS:
Drug: AZD9668 — 20 mg
  Arms: 1; 2
Drug: AZD9668 — 60 mg
  Arms: 3; 4

SUMMARY:
The study is designed to investigate the pharmacokinetic behaviour of the free base formulation of AZD9668. The study will compared the relative bioavailability of the free base formulation at two different dose levels compared to the tosylate salt formulation.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study-specific procedures
* female subjects may be of non-child bearing potential (i.e. post menopausal or surgically sterile).
* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2 calculated from height and weight at the screening visit; minimum weight 50 kg.
* Clinically normal physical and laboratory findings as judged by the investigator, including negative test results for drug-of-abuse, alcohol, cotinine and negative test results for Hepatitis B surface antigen, antibodies to Hepatitis C virus and antibodies to HIV-1/2 at the screening visit
* Be a none smoker or ex-smoker who has stopped smoking for >6 months prior to visit 2 (pre-entry)

Exclusion Criteria:

* Any clinically significant disease or disorder (eg infections/viral disease, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment), which in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the absorption, distribution, metabolism and excretion of drugs.
* Any clinically relevant abnormal findings in physical examination, vital signs, clinical chemistry, haematology, urinalysis, which, in the opinion of the investigator, may put the subject at risk because of his/her participation in the study
* History of cardiac arrhythmia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability (Frel): to assess the relative systemic bioavailability after oral administration of the free base of AZD9668 dosed as a suspension compared to the tosylate salt of AZD9668 dosed as a tablet formulation at two dose levels. | Frequent sampling occasions during the study

SECONDARY OUTCOMES:
Safety variables (adverse events, blood pressure, pulse rate, 12-lead ECG, haematology, clinical chemistry and urinalysis) | Frequent sampling occasions during the study

CONTACTS AND LOCATIONS:
Overall Officials: Emma Harrop, Study Director — AstraZeneca R&D; Rainard Fuhr, Principal Investigator — Parexel
Locations (1):
- Research Site, Berlin, Germany